CLINICAL TRIAL: NCT02875392
Title: Fucoidan Improves the Metabolic Profiles of Patients With Non-alcoholic Fatty Liver Disease (NAFLD)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Taipei Medical University WanFang Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: N201605071
Record Dates: First submitted 2016-08-05; First posted 2016-08-23 (Estimated); Results first posted 2021-03-17 (Actual); Last update posted 2021-04-13 (Actual); Status verified 2016-07

CONDITIONS: Non-alcoholic Fatty Liver Disease
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Fucoidan use (Experimental): FucoHiQ(275mg Oligo Fucoidan + 275mg HS Fucoxanthin) 550mg/capsule 6 per day(before breakfast and supper)
  Interventions: Other: 275mg Oligo Fucoidan + 275mg HS Fucoxanthin
- placebo pills (Placebo Comparator): placebo capsule 6 per day (before breakfast and supper)
  Interventions: Other: placebo pills

INTERVENTIONS:
Other: 275mg Oligo Fucoidan + 275mg HS Fucoxanthin — Fucoidan is a water-soluble dietary fiber which is extracted from brown seaweed. Slimy surface of brown seaweed has unique ingredients and different kind of brown seaweed has slightly different effectiveness.The subject of this study focus on assessing the impact on the metabolism of fatty liver and liver fibrosis after taking oral FucoHiQ capsules.
  Arms: Fucoidan use
Other: placebo pills — taking placebo pills as if patients are under treatment.
  Arms: placebo pills

SUMMARY:
Studies reveal special function of fucoidan so far include anti-virus, anti-tumor, immunomodulatory, anti-inflammatory, blood fat, anti-oxidation and liver and kidney dysfunction and improve fibrosis. The subject of this study focus on assessing the impact on the metabolism of fatty liver and liver fibrosis after taking oral FucoHiQ capsules.

DETAILED DESCRIPTION:
Fucoidan is a water-soluble dietary fiber which is extracted from brown seaweed. Slimy surface of brown seaweed has unique ingredients and different kind of brown seaweed has slightly different effectiveness. The strongest fucoidan among all seaweed for inhibiting cancer cells is in Okinawa Japanese waters. For chemically speaking, the major components for fucoidan consisted of mainly fucose which is a kind of polysaccharide with strong biological activity. However, patients need to take actual fucoidan in order to reach the best effectiveness for inhibiting cancer cell.

Studies reveal special function of fucoidan so far include anti-virus, anti-tumor, immunomodulatory, anti-inflammatory, blood fat, anti-oxidation and liver and kidney dysfunction and improve fibrosis. The subject of this study focus on assessing the impact on the metabolism of fatty liver and liver fibrosis after taking oral FucoHiQ capsules.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are aged between 20-75 with non alcoholic fatty liver disease (NAFLD).

Exclusion Criteria:

1. Patients were allergic to seafood.
2. Patients who take Vitamin E or Pioglitazone.

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2016-11 (Actual); Primary Completion 2017-10 (Actual); Study Completion 2018-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ming-Shung Wu, Doctor, Study Director — Wanfang Hospital
Locations (1):
- WanFangH, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Yang M, Xuan Z, Wang Q, Yan S, Zhou D, Naman CB, Zhang J, He S, Yan X, Cui W. Fucoxanthin has potential for therapeutic efficacy in neurodegenerative disorders by acting on multiple targets. Nutr Neurosci. 2022 Oct;25(10):2167-2180. doi: 10.1080/1028415X.2021.1926140. Epub 2021 May 15. PMID 33993853

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Fucoidan Use | Placebo Pills
Started | 28 | 29
Completed | 21 | 21
Not Completed | 7 | 8
Not completed — The subjects did not inform their Hepatobiliary disorders; hence, their data did not analyze | 7 | 8

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Fucoidan Use | Placebo Pills | Total
Number analyzed (Participants) | 28 | 29 | 57
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 24 | 18 | 42
  >=65 years | 4 | 11 | 15
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 21 | 32
  Male | 17 | 8 | 25
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Change in ALT Index
Description: Measure the first month and the sixth-month change in the index which is ALT related to Liver inflammation.
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | Fucoidan Use | Placebo Pills
Number analyzed (Participants) | 21 | 21
U/L
  First Month | 42.238 (17.196) | 33.524 (21.736)
  Sixth Month | 36.667 (16.01) | 36.238 (22.221)

2. Primary Outcome: Change in AST Index
Description: Measure the first month and the sixth-month change in the index which is AST relate to Liver inflammation
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | Fucoidan Use | Placebo Pills
Number analyzed (Participants) | 21 | 21
U/L
  First Month | 28.095 (7.049) | 27.905 (15.776)
  Sixth Month | 25.286 (7.349) | 28.048 (14.165)

3. Primary Outcome: Change in HbA1c
Description: Measure the first month and the sixth-month change in the index which is HbA1c relate to Liver inflammation
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: percentage of glycated hemoglobin
Arm/Group | Fucoidan Use | Placebo Pills
Number analyzed (Participants) | 21 | 21
percentage of glycated hemoglobin
  First Month | 5.871 (0.443) | 6.057 (0.451)
  Sixth Month | 5.79 (0.525) | 6.152 (0.608)

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Fucoidan Use | Placebo Pills
All-Cause Mortality (participants affected / at risk) | 0/28 | 0/29
Serious Adverse Events (participants affected / at risk) | 0/28 | 0/29
Other Adverse Events (participants affected / at risk) | 0/28 | 0/29

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-07-04): https://cdn.clinicaltrials.gov/large-docs/92/NCT02875392/Prot_SAP_000.pdf